CLINICAL TRIAL: NCT04335682
Title: A Randomized Phase II Study of Androgen Receptor Directed Therapy on COGnitive Function in Patients Treated With Darolutamide or Enzalutamide (ARACOG)
Brief Title: Androgen Receptor Directed Therapy on Cognitive Function in Patients Treated With Darolutamide or Enzalutamide
Acronym: ARACOG
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AFT-47
Record Dates: First submitted 2020-01-13; First posted 2020-04-06 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Prostate Cancer; Prostate Cancer Metastatic; Prostate Cancer; Castrate Resistant Prostate Cancer; Hormone Sensitive Prostate Cancer; Non-metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Darolutamide (DARO) (Active Comparator): Patients will take DARO at a dose of 600 mg (300 mg ×2 tablets) by mouth twice daily beginning on Day 1, of Week 1. Patients will take DARO throughout planned treatment period or withdrawal of consent or progression of disease requiring change in therapy.
  Interventions: Drug: Darolutamide
- Enzalutamide (ENZ) (Active Comparator): Patients will take ENZ at a dose of 160 mg PO once daily (QD), beginning on Day 1, of Week 1. Patients will take ENZ throughout planned treatment period or withdrawal of consent or progression of disease requiring change in therapy.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Darolutamide — Patients randomized to darolutamide.
  Other Names: Nubeqa
  Arms: Darolutamide (DARO)
Drug: Enzalutamide — Patients randomized to enzalutamide.
  Other Names: Xtandi
  Arms: Enzalutamide (ENZ)

SUMMARY:
This is a prospective, randomized, open-label phase II study comparing cognitive outcomes between men with metastatic and non-metastatic castration resistant prostate cancer (CRPC) or metastatic hormone sensitive prostate cancer (HSPC). Approximately 132 patients will be enrolled. Eligible patients will be randomized in a 1:1 fashion to treatment with enzalutamide 160 mg orally daily or darolutamide 600 mg orally twice daily, in combination with standard LHRH agonist based treatment. Cognitive assessments will be performed using modules from Cambridge Neuropsychological Test Automated Battery (CANTAB) an internationally recognized software for assessing cognitive function and impairment.

DETAILED DESCRIPTION:
The goal of the trial is to assess cognitive and quality of life outcomes over the 48-week primary data collection period of the trial. This is a prospective, randomized, open-label phase II study comparing cognitive outcomes between men with Advanced prostate cancer: metastatic and non-metastatic castration resistant prostate cancer (CRPC) or metastatic hormone sensitive prostate cancer (HSPC).

The primary endpoint will be the percent change in the maximally changed cognitive domain by 24 weeks in each study arm. Patients will be stratified by age (<65, 65-80, > 80). Patients will be allowed to cross over from either treatment to the opposite treatment arm at 12 and 24 weeks if they meet any of the cross-over criteria as described in the protocol.

Cognitive assessments will be performed using Cambridge Neuropsychological Test Automated Battery (CANTAB), an internationally recognized software for assessing cognitive function and impairment. Tests available in the CANTAB battery include tests of learning and executive function; working memory; visual, verbal and episodic memory; and attention, information and processing time. The maximally changed cognitive domain is defined as the domain most changed from baseline in each individual.

Blood samples will be collected for exploratory genomic analyses (AR CAG repeat length, PHS, exosome analysis).

Patients will have the option to opt into an additional separate MRI sub-study. A subset of 40 patients (20 per arm) will undergo fMRI to measure percent signal change in the HP PFC circuit at baseline, 24 and 48 weeks or/and cross-over/end of treatment visit (if applicable).

ELIGIBILITY:
Key inclusion criteria include:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Progressive disease per PCWG3 criteria with EITHER: Metastatic CRPC or non- metastatic CRPC (M0CRPC)

  * For mCRPC: metastatic disease documented by standard or novel imaging techniques
  * OR for M0CPRC: no evidence of metastatic disease on standard imaging.
* OR mHSPC
* Surgically or medically castrated, with testosterone levels of <50 ng/dL. If the patient is medically castrated, continuous dosing with GnRH agonist or antagonist must have been initiated at least 4 weeks prior to randomization and must be continued throughout the study.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Able to complete cognitive testing and patient reported outcome surveys in English.
* Ability to swallow study medications whole.
* Able to provide informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in the maximally changed cognitive domain | 24 weeks
  To compare the effects of treatment with enzalutamide (ENZ) versus darolutamide (DARO) on the cognitive function of men with non-metastatic and metastatic castration-resistant prostate cancer by comparing the change in the maximally changed cognitive domain utilizing Cambridge Neuropsychological Test Automated Battery [CANTAB] cognitive tests from baseline in patients in each study arm.Tests available in the CANTAB battery include tests of learning and executive function; working memory; visual, verbal and episodic memory; and attention, information and processing time. The maximally changed cognitive domain is defined as the domain most changed from baseline in each individual.

SECONDARY OUTCOMES:
Crossover from enzalutamide to darolutamide and darolutamide to enzalutamide | 48 weeks
  Proportion of patients crossing over from each treatment arm based on subjective (self-reported, FACT-Cognitive Function [Version 3], FACT-Cog V3, decline by >10 points from baseline score) cognitive effects.
  * Proportion of patients crossing over from each treatment arm based on objective cognitive effects (the Cambridge Neuropsychological Test Automated Battery [CANTAB] , decline by > 30% from baseline on any cognitive domain).
  * Proportion of patients crossing over from ENZ to DARO based on Timed Up and Go (TUG) times >12 seconds or 12 seconds or increase from baseline by >1 second.
  * Proportion of patient crossing over due to neurologic toxicity (fatigue) with a preference to cross over (ENZ or DARO) or severe neurological toxicity [seizures or posterior reversible encephalopathy syndrome PRES]). Cross over for severe neurologic toxicity is allowed for patients on ENZ only.
Maximally changed cognitive domain | 48 weeks
  Average decline in maximally changed cognitive domain in patients in each arm based on self-reported cognitive tests (Cambridge Neuropsychological Test Automated Battery [CANTAB]). Tests in the CANTAB battery include tests of learning and executive function; working memory; visual, verbal and episodic memory; and attention, information and processing time. The maximally changed cognitive domain is defined as the domain most changed from baseline in each individual.
Proportion of impaired patients | 24 weeks
  Cumulative proportion of impaired patients in each arm
Proportion of impaired patients | 48 weeks
  Cumulative proportion of impaired patients in each arm
Change in lowest ranking domain | 24 weeks
  Average change in lowest ranking domain Cambridge Neuropsychological Test Automated Battery [CANTAB] questionnaire outcomes at baseline (in a given individual). Tests in the CANTAB battery include tests of learning and executive function; working memory; visual, verbal and episodic memory; and attention, information and processing time.
Change in lowest ranking domain | 48 weeks
  Average change in lowest ranking domain in Cambridge Neuropsychological Test Automated Battery [CANTAB] outcomes at baseline (in a given individual). Tests in the CANTAB battery include tests of learning and executive function; working memory; visual, verbal and episodic memory; and attention, information and processing time.
Improve in cognitive function after crossover | 48 weeks
  Improvement in cognitive function after crossover from each treatment arm based on Cambridge Neuropsychological Test Automated Battery [CANTAB] modules. Tests in the CANTAB battery include tests of learning and executive function; working memory; visual, verbal and episodic memory; and attention, information and processing time.
Prostate-specific antigen (PSA) progression. | 104 weeks
  Estimation of the probability of PSA progression over time using the cumulative incidence function.
Progression free survival | 104 weeks
  Progression-free survival will be evaluated for each cohort.
Prostate-specific antigen (PSA) response rate | 24 weeks
  Estimation or the proportion PSA responses at 24 weeks (on the basis of a decrease from baseline of ≥ 50%)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, MD, Principal Investigator — Alliance Foundation Trials
Locations (8):
- United States (8):
  - University of California - San Francisco at Mount Zion, San Francisco, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Kansas Cancer Center, Fairway, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Fizazi K, Shore N, Tammela TL, Ulys A, Vjaters E, Polyakov S, Jievaltas M, Luz M, Alekseev B, Kuss I, Kappeler C, Snapir A, Sarapohja T, Smith MR; ARAMIS Investigators. Darolutamide in Nonmetastatic, Castration-Resistant Prostate Cancer. N Engl J Med. 2019 Mar 28;380(13):1235-1246. doi: 10.1056/NEJMoa1815671. Epub 2019 Feb 14. PMID 30763142
- [Background] Apple AC, Ryals AJ, Alpert KI, Wagner LI, Shih PA, Dokucu M, Cella D, Penedo FJ, Voss JL, Wang L. Subtle hippocampal deformities in breast cancer survivors with reduced episodic memory and self-reported cognitive concerns. Neuroimage Clin. 2017 Mar 16;14:685-691. doi: 10.1016/j.nicl.2017.03.004. eCollection 2017. PMID 28377882
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Wang L, Apple AC, Schroeder MP, Ryals AJ, Voss JL, Gitelman D, Sweet JJ, Butt ZA, Cella D, Wagner LI. Reduced prefrontal activation during working and long-term memory tasks and impaired patient-reported cognition among cancer survivors postchemotherapy compared with healthy controls. Cancer. 2016 Jan 15;122(2):258-68. doi: 10.1002/cncr.29737. Epub 2015 Oct 20. PMID 26484435
- [Background] de Souza JA, Yap BJ, Wroblewski K, Blinder V, Araujo FS, Hlubocky FJ, Nicholas LH, O'Connor JM, Brockstein B, Ratain MJ, Daugherty CK, Cella D. Measuring financial toxicity as a clinically relevant patient-reported outcome: The validation of the COmprehensive Score for financial Toxicity (COST). Cancer. 2017 Feb 1;123(3):476-484. doi: 10.1002/cncr.30369. Epub 2016 Oct 7. PMID 27716900
- [Background] Hussain M, Fizazi K, Saad F, Rathenborg P, Shore N, Ferreira U, Ivashchenko P, Demirhan E, Modelska K, Phung D, Krivoshik A, Sternberg CN. Enzalutamide in Men with Nonmetastatic, Castration-Resistant Prostate Cancer. N Engl J Med. 2018 Jun 28;378(26):2465-2474. doi: 10.1056/NEJMoa1800536. PMID 29949494
- [Background] Evans CP, Higano CS, Keane T, Andriole G, Saad F, Iversen P, Miller K, Kim CS, Kimura G, Armstrong AJ, Sternberg CN, Loriot Y, de Bono J, Noonberg SB, Mansbach H, Bhattacharya S, Perabo F, Beer TM, Tombal B. The PREVAIL Study: Primary Outcomes by Site and Extent of Baseline Disease for Enzalutamide-treated Men with Chemotherapy-naive Metastatic Castration-resistant Prostate Cancer. Eur Urol. 2016 Oct;70(4):675-683. doi: 10.1016/j.eururo.2016.03.017. Epub 2016 Mar 19. PMID 27006332
- [Background] Lim YY, Pietrzak RH, Ellis KA, Jaeger J, Harrington K, Ashwood T, Szoeke C, Martins RN, Bush AI, Masters CL, Rowe CC, Villemagne VL, Ames D, Darby D, Maruff P. Rapid decline in episodic memory in healthy older adults with high amyloid-beta. J Alzheimers Dis. 2013;33(3):675-9. doi: 10.3233/JAD-2012-121516. PMID 23001710
- [Background] Rosario ER, Carroll JC, Pike CJ. Evaluation of the effects of testosterone and luteinizing hormone on regulation of beta-amyloid in male 3xTg-AD mice. Brain Res. 2012 Jul 23;1466:137-45. doi: 10.1016/j.brainres.2012.05.011. Epub 2012 May 14. PMID 22587890
- [Background] Cherrier MM, Aubin S, Higano CS. Cognitive and mood changes in men undergoing intermittent combined androgen blockade for non-metastatic prostate cancer. Psychooncology. 2009 Mar;18(3):237-47. doi: 10.1002/pon.1401. PMID 18636420
- [Background] Nead KT, Gaskin G, Chester C, Swisher-McClure S, Leeper NJ, Shah NH. Association Between Androgen Deprivation Therapy and Risk of Dementia. JAMA Oncol. 2017 Jan 1;3(1):49-55. doi: 10.1001/jamaoncol.2016.3662. PMID 27737437
- [Background] Gonzalez BD, Jim HS, Booth-Jones M, Small BJ, Sutton SK, Lin HY, Park JY, Spiess PE, Fishman MN, Jacobsen PB. Course and Predictors of Cognitive Function in Patients With Prostate Cancer Receiving Androgen-Deprivation Therapy: A Controlled Comparison. J Clin Oncol. 2015 Jun 20;33(18):2021-7. doi: 10.1200/JCO.2014.60.1963. Epub 2015 May 11. PMID 25964245